CLINICAL TRIAL: NCT05817123
Title: Psychometric Validation of the Mutuality Scale in Patients With Obstructive Sleep Apnea and Their Partners
Brief Title: Validation of the Mutuality Scale in Patients With OSA and Their Partners
Acronym: VAMOS
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09C123
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSAS patients: Patients with Obstructive Sleep Apnea Syndrome
  Interventions: Other: Questionnaires
- Partners: Partners of OSAS patients
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Administration of the following questionnaires:
  * Mutuality scale
  * Pittsburgh Sleep Quality Index (PSQI)
  * Epworth Sleep Scale (ESS)
  * Sleep Condition Indicator (SCI)
  * International Physical Activity Questionaire (IPAQ)
  * Mediterranean diet score (MDS)
  * Quality of Life SF 12
  * Hospital Anxiety and Depression Scale (HADS)

SUMMARY:
Main objective of this study is to assess the psychometric characteristics of the Mutuality Scale both in patients with Obstructive Sleep Apnea Syndrome (OSAS) and in their partners-The association between the mutuality score in OSAS patients and their adherence to the use of Continuous Positive Airway Pressure (CPAP) therapy will also be investigated.

The results of the study may allow a validation of the Mutuality Score as an instrument for measuring mutuality between OSAS patients and their partners.

ELIGIBILITY:
OSA patients:

Inclusion Criteria:

* Age 18 years and older

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Obstructive Sleep Apnea Syndrome (OSAS) and their partners
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Score on Mutuality Scale in OSAS patients | At baseline
  15-item scale; points for every item 0-4; minimum score 0; maximum score 60
Score on Mutuality Scale in partners | At baseline
  15-item scale; points for every item 0-4; minimum score 0; maximum score 60

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy